CLINICAL TRIAL: NCT00551330
Title: Vicriviroc in Combination Treatment With an Optimized ART Regimen in Treatment-Experienced Subjects With R5/X4 HIV Infection (VICTOR-E2; Protocol No. P05057)
Brief Title: Vicriviroc in HIV(R5/X4)-Treatment Experienced Subjects (Study P05057AM5)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05057
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: HIV Infections; Acquired Immunodeficiency Syndrome
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — vicriviroc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Vicriviroc 30 mg QD
  Interventions: Drug: Vicriviroc
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vicriviroc — One tablet of vicriviroc 30 mg once daily
  Arms: 1
Drug: Placebo — One tablet of placebo once daily
  Arms: 2

SUMMARY:
Vicriviroc (vye-kri-VYE-rock) is an investigational drug (not yet approved by Government Regulatory Authorities for commercial use) that belongs to a new class of drugs, called CCR5 receptor blockers. This group of drugs blocks one of the ways HIV enters T-cells (the cells that fight infection). Previous smaller studies in HIV treatment-experienced patients, have shown that vicriviroc is safe and effective. The purpose of this study is to investigate in subjects with detectable dual/mixed CCR5/CXCR4-tropic HIV whether vicriviroc when added to other appropriate HIV drugs can decrease the level of HIV (viral load) in the blood and that it is well tolerated.

This is a randomized, double-blind, placebo-controlled, parallel-group, multi-center study of vicriviroc maleate in HIV subjects infected with dual/mixed CCR5/CXCR4-tropic virus and who have documented resistance to at least 2 of the 3 antiretroviral drug classes (NRTI, NNRTI or PI) or at least 6 months experience with at least 2 of the following: one NRTI, one NNRTI, or one PI (excluding low-dose ritonavir) and failure on their current stable regimen. The study will compare the virologic benefit of adding vicriviroc to an optimized background regimen to a control group receiving placebo plus the new optimized background therapy. The optimized background regimen will be chosen by the investigator based on results of drug susceptibility tests performed at Screening, history of prior antiretroviral drug use by the patient, and drug toxicity. Primary efficacy analysis will be conducted when all subjects have completed 48 weeks of treatment. An interim analysis will be performed when all subjects have completed 24 weeks of treatment. Subjects who complete 48 weeks of treatment, or who discontinue early but are deemed eligible upon rescreening, will be offered participation in the open-label segment of the study, and will receive vicriviroc 30 mg once daily, if appropriate, until commercially available or until the sponsor terminates the clinical development of vicriviroc.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 16 years of age (or minimal age that defines an adult as determined by local regulatory authorities or legal requirements), of either sex and of any race, with dual/mixed CCR5/CXCR4 tropic HIV infection.
* Subjects must have treatment failure (defined by plasma HIV RNA [ribonucleic acid] >1000 copies/mL) on an existing regimen.
* Subjects must be antiretroviral therapy (ART)-experienced and have documented genotypic and/or phenotypic resistance to at least one drug in 2 of the following 3 drug classes: nucleoside reverse transcriptase inhibitor (NRTI), nonnucleoside reverse transcriptase inhibitor (NNRTI), or protease inhibitor (PI)

OR

* Antiretroviral class experience for at least 6 months (sequential or cumulative) with at least two of the following:

  * one NRTI
  * one NNRTI
  * one PI (excluding low dose ritonavir).
* In the opinion of the investigator, the best treatment regimen for the subject must be an optimized ART regimen consisting of >=3 drugs, the optimized regimen must contain at least 2 active drugs, one of which must be a ritonavir-boosted PI (>=100 mg ritonavir). With the exception of etravirine, NNRTIs may not be a component of the optimized regimen.

Exclusion Criteria:

* Any condition likely to increase the risk of seizures.
* CD4 count <100 cells/mm^3.
* Current or prior history of malignancy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2007-09; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HIV RNA (log10 copies/mL) | At Week 48

SECONDARY OUTCOMES:
Change from baseline in CD4 count | At Week 24 and Week 48